CLINICAL TRIAL: NCT03686033
Title: A Multicenter, Double-Blind, Randomized, Crossover, Single-Dose Study With An Open-Label Treatment Period Evaluating Pharmacodynamic Activity of E2082 in Adult Subjects With Photosensitive Epilepsy
Brief Title: A Study to Evaluate the Pharmacodynamic Activity of E2082 in Adult Participants With Photosensitive Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety Review
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2082-A001-201
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2018-08

CONDITIONS: Photosensitive Epilepsy
Keywords: E2082; Epilepsy; Photosensitive; Anti-epileptic; Seizures; Photoparoxysmal response; PPR
MeSH Terms: conditions — Epilepsy, Reflex; Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: The study consists of a crossover design in Treatment Periods 1, 2, and 3, followed by an open-label Treatment Period 4.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study consists of a randomized double-blind design in Treatment Periods 1, 2, and 3, followed by an open-label Treatment Period 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo, E2082 2.5 mg, E2082 25 mg, E2082 40 mg (Experimental): Participants will receive a single dose of E2082-matched placebo tablet orally (Treatment A) in Treatment Period 1 followed by a single dose of E2082 tablets at 2.5 mg orally (Treatment B) in Treatment Period 2 followed by a single dose of E2082 tablets at 25 mg orally (Treatment C) in Treatment Period 3 followed by a single dose of E2082 tablets at 40 mg orally in Treatment Period 4. A wash-out phase of at least 2 weeks will be maintained between all the treatment periods.
  Interventions: Drug: Placebo; Drug: E2082
- E2082 2.5 mg, E2082 25 mg, Placebo, E2082 40 mg (Experimental): Participants will receive a single dose of E2082 tablets at 2.5 mg orally (Treatment B) in Treatment Period 1 followed by a single dose of E2082 tablets at 25 mg orally (Treatment C) in Treatment Period 2 followed by a single dose of E2082-matched placebo tablet orally (Treatment A) in Treatment Period 3 followed by a single dose of E2082 tablets at 40 mg orally in Treatment Period 4. A wash-out phase of at least 2 weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2082
- E2082 25 mg, Placebo, E2082 2.5 mg, E2082 40 mg (Experimental): Participants will receive a single dose of E2082 tablets at 25 mg orally (Treatment C) in Treatment Period 1 followed by a single dose of E2082-matched placebo tablet orally (Treatment A) in Treatment Period 2 followed by a single dose of E2082 tablets at 2.5 mg orally (Treatment B) in Treatment Period 3 followed by a single dose of E2082 tablets at 40 mg orally in Treatment Period 4. A wash-out phase of at least 2 weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2082
- Placebo, E2082 25 mg, E2082 2.5 mg, E2082 40 mg (Experimental): Participants will receive a single dose of E2082-matched placebo tablet orally (Treatment A) in Treatment Period 1 followed by a single dose of E2082 tablets at 25 mg orally (Treatment C) in Treatment Period 2 followed by a single dose of E2082 tablets at 2.5 mg orally (Treatment B) in Treatment Period 3 followed by a single dose of E2082 tablets at 40 mg orally in Treatment Period 4. A wash-out phase of at least 2 weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2082
- E2082 2.5 mg, Placebo, E2082 25 mg, E2082 40 mg (Experimental): Participants will receive a single dose of E2082 tablets at 2.5 mg orally (Treatment B) in Treatment Period 1 followed by a single dose of E2082-matched placebo tablet orally (Treatment A) in Treatment Period 2 followed by a single dose of E2082 tablets at 25 mg orally (Treatment C) in Treatment Period 3 followed by a single dose of E2082 tablets at 40 mg orally in Treatment Period 4. A wash-out phase of at least 2 weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2082
- E2082 25 mg, E2082 2.5 mg, Placebo, E2082 40 mg (Experimental): Participants will receive a single dose of E2082 tablets at 25 mg orally (Treatment C) in Treatment Period 1 followed by a single dose of E2082 tablets at 2.5 mg orally (Treatment B) in Treatment Period 2 followed by a single dose of E2082-matched placebo tablet orally (Treatment A) in Treatment Period 3 followed by a single dose of E2082 tablets at 40 mg orally in Treatment Period 4. A wash-out phase of at least 2 weeks will be maintained between the treatment periods.
  Interventions: Drug: Placebo; Drug: E2082

INTERVENTIONS:
Drug: Placebo — Participants will receive E2082-matched placebo tablets orally.
Drug: E2082 — Participants will receive E2082 tablets orally.

SUMMARY:
The primary purpose of the study is to assess pharmacodynamic (PD) activity of E2082 as measured by suppression of epileptic photoparoxysmal response (PPR) in the participant's most sensitive eye condition in participants with photosensitive epilepsy, compared to placebo.

ELIGIBILITY:
1. Diagnosis and/or history of a PPR on EEG.
2. If currently being treated with antiepileptic drug (AED), up to a maximum of 3 concomitant AEDs is allowed provided that doses must have remained stable for at least 4 weeks (or at least 8 weeks if recently initiated) before screening.
3. Reproducible IPS-induced PPR on EEG of at least 3 points on the SPR scale in at least 1 eye condition (eye closure, eyes closed, eyes open) on at least 3 of the EEGs performed at screening.
4. Body mass index (BMI) between 18 to 35 kilogram per square meter (kg/m^2) (inclusive) and a total body weight greater than or equal to (>=) 45 kilogram (kg) at screening.
5. Agrees to refrain from strenuous exercise and alcohol consumption during the 24-hour period before screening and before each treatment day.

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at screening or baseline.
2. Male participants who have not had a successful vasectomy, they and their female partners not of childbearing potential, or practicing highly effective contraception throughout the study period and for 28 days after study drug discontinuation. No sperm donation is allowed during the study period and for 28 days after study drug discontinuation.
3. History of nonepileptic seizures (example, metabolic, structural, or pseudoseizures) while on any antiepileptic medication.
4. History of status epilepticus while on any antiepileptic medication(s) within 2 years before screening.
5. Ongoing or history of generalized tonic-clonic seizures (GTCS) within 6 months before screening.
6. Participants who had developed a clinical seizure during previous PPR assessment, or who experiences a clinical seizure during the Screening IPS procedure.
7. Frequent spontaneous background burst or current evidence of proconvulsive activity on EEG (example, increase in spike-wave activity) at screening.
8. Inability to follow restriction on watching television, or use of any device(s) with an animated screen (example, computer, video games, tablets, or smart phone) from the time of arrival at the study center until study procedures are completed for that day.
9. Use of perampanel within 6 weeks before screening.
10. Use of felbamate for less than 2 years or where the dose has not been stable for at least 8 weeks before Visit 1.
11. Use of vigabatrin within 5 months before screening and/or documented evidence of vigabatrin associated clinically significant abnormality in a visual perimetry test.
12. Use of benzodiazepines for non-epilepsy related indications. Intermittent use of benzodiazepines as rescue medication or stable dosage (greater than 4 weeks before screening) for epilepsy indications is allowed.
13. Concomitant use of cannabinoids.
14. Use of concomitant potent cytochrome P450 (CYP)3A inducers or inhibitors within 4 weeks or 5 half-lives, whichever is longer.
15. Vagus nerve stimulation (VNS) implanted within 5 months or changes in parameter within 4 weeks before screening.
16. On a ketogenic diet for which the diet is not a stable regimen for at least 4 weeks before screening.
17. Participants with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
18. A history of prolonged QT syndrome or risk factors for torsade de pointes, or the use of concomitant medications that cause QT prolongation as demonstrated on screening electrocardiogram (ECG).
19. Any suicidal ideation with intent with or without a plan within 6 months before or during screening, and/or any lifetime suicidal behavior.
20. Any psychotic disorder(s) or unstable recurrent affective disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Clinical Trials, Inc. and Arkansas Epilepsy Program, Little Rock, Arkansas
  - Consultants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Johns Hopkins University- School of Medicine, Baltimore, Maryland
  - Washington University Hospital, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 31 October 2018 to 18 June 2019. A total of 8 participants were screened and enrolled, of which 5 participants were randomized and treated, of which, 4 participants completed both crossover and open label treatments in the study.
Pre-assignment Details: The study was terminated due to safety concerns from a phase 1 study (E2082-J081-001; NCT03402178) and preclinical animal toxicity testing.
Groups:
- Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg: Participants received, E2082-matched placebo (Treatment A) tablet, orally, once on Day 1 in Treatment Period 1, followed by E2082 2.5 milligram (mg) (Treatment B) tablet, orally, once on Day 1 in Treatment Period 2, followed by E2082 25 mg (Treatment C) tablet, orally, once on Day 1 in Treatment Period 3, followed by E2082 40 mg tablet, orally, once on Day 1 in Treatment Period 4 (Open-label). A washout phase of at least 2 weeks was maintained between all the treatment periods.
- Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg: Participants received, E2082 2.5 mg (Treatment B) tablet, orally, once on Day 1 in Treatment Period 1, followed by E2082 25 mg (Treatment C) tablet, orally, once on Day 1 in Treatment Period 2, followed by E2082-matched placebo (Treatment A) tablet, orally, once on Day 1 in Treatment Period 3, followed by E2082 40 mg tablet, orally, once on Day 1 in Treatment Period 4 (Open-label). A washout phase of at least 2 weeks was maintained between the treatment periods.
- Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg: Participants received, E2082 25 mg (Treatment C) tablet, orally, once on Day 1 in Treatment Period 1, followed by E2082-matched placebo (Treatment A) tablet, orally, once on Day 1 in Treatment Period 2, followed by E2082 2.5 mg (Treatment B) tablet, orally, once on Day 1 in Treatment Period 3, followed by E2082 40 mg tablet, orally, once on Day 1 in Treatment Period 4 (Open-label). A washout phase of at least 2 weeks was maintained between the treatment periods.
- Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg: Participants received, E2082-matched placebo (Treatment A) tablet, orally, once on Day 1 in Treatment Period 1, followed by E2082 25 mg (Treatment C) tablet, orally, once on Day 1 in Treatment Period 2, followed by E2082 2.5 mg (Treatment B) tablet, orally, once on Day 1 in Treatment Period 3, followed by E2082 40 mg tablet, orally, once on Day 1 in Treatment Period 4 (Open-label). A washout phase of at least 2 weeks was maintained between the treatment periods.
- Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg: Participants received, E2082 2.5 mg (Treatment B) tablet, orally, once on Day 1 in Treatment Period 1, followed by E2082-matched placebo (Treatment A) tablet, orally, once on Day 1 in Treatment Period 2, followed by E2082 25 mg (Treatment C) tablet, orally, once on Day 1 in Treatment Period 3, followed by E2082 40 mg tablet, orally, once on Day 1 in Treatment Period 4 (Open-label). A washout phase of at least 2 weeks was maintained between the treatment periods.
- Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg: Participants received, E2082 25 mg (Treatment C) tablet, orally, once on Day 1 in Treatment Period 1, followed by E2082 2.5 mg (Treatment B) tablet, orally, once on Day 1 in Treatment Period 2, followed by E2082-matched placebo (Treatment A) tablet, orally, once on Day 1 in Treatment Period 3, followed by E2082 40 mg tablet, orally, once on Day 1 in Treatment Period 4 (Open-label). A washout phase of at least 2 weeks was maintained between the treatment periods.
Period: Treatment Period 1 (1 Day)
Arm/Group | Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg | Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg | Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg | Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg | Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg | Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg
Started | 1 | 1 | 1 | 1 | 1 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Phase (at Least 2 Weeks)
Arm/Group | Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg | Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg | Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg | Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg | Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg | Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg
Started | 1 | 1 | 1 | 1 | 1 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (1 Day)
Arm/Group | Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg | Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg | Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg | Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg | Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg | Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg
Started | 1 | 1 | 1 | 1 | 1 | 0
Completed | 1 | 1 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Phase (at Least 2 Weeks)
Arm/Group | Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg | Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg | Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg | Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg | Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg | Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg
Started | 1 | 1 | 1 | 1 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (1 Day)
Arm/Group | Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg | Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg | Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg | Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg | Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg | Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg
Started | 1 | 1 | 1 | 1 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Phase (at Least 2 Weeks)
Arm/Group | Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg | Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg | Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg | Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg | Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg | Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg
Started | 1 | 1 | 1 | 1 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4 (1 Day)
Arm/Group | Sequence 1: Placebo + E2082 2.5 mg + E2082 25 mg + E2082 40 mg | Sequence 2: E2082 2.5 mg + E2082 25 mg + Placebo + E2082 40 mg | Sequence 3: E2082 25 mg + Placebo + E2082 2.5 mg + E2082 40 mg | Sequence 4: Placebo + E2082 25 mg + E2082 2.5 mg + E2082 40 mg | Sequence 5: E2082 2.5 mg + Placebo + E2082 25 mg + E2082 40 mg | Sequence 6: E2082 25 mg + E2082 2.5 mg + Placebo + E2082 40 mg
Started | 1 | 1 | 1 | 1 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug and have at least 1 postdose safety assessment.
Groups:
- Overall Participants: Participants received E2082-matched placebo (Treatment A) or E2082 2.5 mg (Treatment B) or E2082 25 mg (Treatment C) and E2082 40 mg tablet, orally, once on Day 1 in Treatment Period 1 to 4 as per assigned treatment sequence. A washout phase of at least 2 weeks was maintained between all the treatment periods.
Arm/Group | Overall Participants
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 60 years | 5
  >=60 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Photoparoxysmal Response (PPR) Range in the Most Sensitive Eye Condition at 8 Hours Postdose on Day 1 of Each Treatment Period
Description: PPR was an electroencephalogram (EEG) trait of spike and spike-wave discharges in response to photic stimulation. Intermittent photic stimulation (IPS)-EEG assessments determine the range of frequencies of IPS that elicited an epileptiform EEG response. Each IPS-EEG assessment was conducted in all 3 eye conditions (eye closure, eyes closed, and eyes open) at ascending and then descending photo stimulation administered at 14 standard frequencies: 2, 5, 8, 10, 13, 15, 18, 20, 23, 25, 30, 40, 50, and 60 hertz (Hz). The lower and upper limit of photosensitivity to IPS threshold frequency were determined for each eye condition. From this range, standard photosensitivity response (SPR) was derived. SPR is an integer score that ranges from 0 to 14, with lower scores representing better outcomes. Most sensitive eye condition was defined as one that yielded the largest SPR before dosing.
Time Frame: Baseline (30 minutes-2 hours) and at 8 hours postdose on Day 1 of each treatment period
Population: The pharmacodynamic (PD) analysis set was the group of randomized participants who received at least 1 dose of study drug and have sufficient PD data to derive at least 1 PD parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment A: Placebo: Participants received, E2082-matched placebo tablet, orally, once on Day 1 as per assigned Treatment sequence in Treatment Period 1, 2, or 3.
- Treatment B: E2082 2.5 mg: Participants received, E2082 2.5 mg tablet, orally, once on Day 1 as per assigned treatment sequence in Treatment Period 1, 2, or 3.
- Treatment C: E2082 25 mg: Participants received, E2082 25 mg tablet, orally, once on Day 1 as per assigned treatment sequence in Treatment Period 1, 2, or 3.
- Open-label Treatment: E2082 40 mg: Participants received, E2082 40 mg, tablet, orally, once on Day 1 of Treatment Period 4 in all the sequences.
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
units on a scale
  Baseline | 6.80 (4.604) | 5.60 (4.336) | 6.00 (3.651) | 6.50 (1.732)
  Change at 8 hours postdose | 0.00 (1.517) | 1.16 (1.381) | -3.90 (2.928) | -5.25 (0.957)
Statistical Analysis 1: Comparison: Treatment A: Placebo vs Treatment B: E2082 2.5 mg; The mixed effects model for the crossover part of the study will include treatment, period, and sequence as fixed effects, baseline (predose) measurement as a covariate, and subject nested within sequence as a random effect. Least Square (LS) Mean Difference was calculated for 2.5 mg versus (vs) Placebo only; Test type: Superiority; LS Mean difference = 1.12, 90% CI 2-sided [-0.98 to 3.22]
Statistical Analysis 2: Comparison: Treatment A: Placebo vs Treatment C: E2082 25 mg; The mixed effects model for the crossover part of the study will include treatment, period, and sequence as fixed effects, baseline (predose) measurement as a covariate, and subject nested within sequence as a random effect. LS Mean Difference was calculated for 25 mg vs Placebo only; Test type: Superiority; LS Mean difference = -4.17, 90% CI 2-sided [-6.35 to -1.99]

2. Secondary Outcome: Mean Change From Baseline in PPR Ranges in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Opened) at 8 Hours Postdose on Day 1 of Each Treatment Period
Description: PPR was an EEG trait of spike and spike-wave discharges in response to photic stimulation. IPS-EEG assessments determine the range of frequencies of IPS that elicited an epileptiform EEG response. Each IPS-EEG assessment was conducted in all 3 eye conditions (eye closure, eyes closed, and eyes open) at ascending and then descending photo stimulation administered at 14 standard frequencies: 2, 5, 8, 10, 13, 15, 18, 20, 23, 25, 30, 40, 50, and 60 Hz. The lower and upper limit of photosensitivity to IPS threshold frequency were determined for each eye condition. From this range, SPR was derived. SPR is an integer score that ranges from 0 to 14, with lower scores representing better outcomes.
Time Frame: Baseline (30 minutes-2 hours) and at 8 hours postdose on Day 1 of each treatment period
Population: The PD analysis set was the group of randomized participants who received at least 1 dose of study drug and have sufficient PD data to derive at least 1 PD parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-label Treatment: E2082 40 mg: Participants received, E2082 40 mg tablet, orally, once on Day 1 of Treatment Period 4 in all the sequences.
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
units on a scale
  Eye Closure: Baseline | 6.2 (4.09) | 6 (3.87) | 5.8 (4.65) | 5.5 (2.89)
  Eye Closure: Change at 8 hours postdose | 0.6 (1.66) | 0.4 (0.91) | -3.7 (3.93) | -4.3 (1.71)
  Eyes Closed: Baseline | 5.4 (4.72) | 5.6 (4.72) | 5.3 (3.2) | 6.3 (2.87)
  Eyes Closed: Change at 8 hours postdose | 1.1 (1.4) | 0.7 (1.56) | -3.7 (2.96) | -5.4 (1.62)
  Eyes Open: Baseline | 5.2 (5.4) | 4.6 (4.04) | 5 (3.83) | 6.3 (4.65)
  Eyes Open: Change at 8 hours postdose | 0.5 (2.18) | 0.8 (1.12) | -3.9 (3.28) | -5.8 (4.09)

3. Secondary Outcome: Time to Onset of Mean Photosensitivity Response in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Open Condition) up to 8 Hours Postdose on Day 1 of Each Treatment Period
Description: Time to onset of mean photosensitivity response in each of the 3 eye conditions (eye closure, eyes closed, and eyes open condition) was determined from mean and mean change from baseline SPR data across participants. The onset of mean suppression was defined as the first time point at which the mean Response of standardized photosensitivity response (SPR) across participants (not for each participant) was at least 3 units below the mean SPR at baseline. Photosensitivity response were essentially intermittent photosensitivity (intermittent photic stimulation [IPS]) assessments, is a form of visual stimulation, when the participants are flashed with light on their eyes intermittently at different hertz.
Time Frame: Baseline (30 minutes-2 hours) up to 8 hours postdose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Number; unit: hours
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
hours
  Eye Closure | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | 1 | 1
  Eyes Closed | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | 1 | 1
  Eyes Opened | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Time to onset of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | 1 | 1

4. Secondary Outcome: Maximum Change From Baseline of Photosensitivity Response in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Open Condition) up to 8 Hours Postdose on Day 1 of Each Treatment Period
Description: Maximum change from baseline of photosensitivity response in each of the 3 eye conditions (eye closure, eyes closed, and eyes open condition) were reported. PPR was an EEG trait of spike and spike-wave discharges in response to photic stimulation. IPS-EEG assessments determine the range of frequencies of IPS that elicited an epileptiform EEG response. Each IPS-EEG assessment was conducted in all 3 eye conditions (eye closure, eyes closed, and eyes open) at ascending and then descending photo stimulation administered at 14 standard frequencies: 2, 5, 8, 10, 13, 15, 18, 20, 23, 25, 30, 40, 50, and 60 Hz. The lower and upper limit of photosensitivity to IPS threshold frequency were determined for each eye condition. From this range, SPR was derived. SPR is an integer score that ranges from 0 to 14, with lower scores representing better outcomes.
Time Frame: Baseline (30 minutes-2 hours) up to 8 hours postdose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
units on a scale
  Eye Closure: Baseline | 6.20 (4.087) | 6.00 (3.873) | 5.75 (4.646) | 5.50 (2.887)
  Eye Closure: Maximum Change | 1.40 (3.912) | 1.80 (2.588) | -4.50 (3.697) | -5.25 (2.500)
  Eyes Closed: Baseline | 5.40 (4.722) | 5.60 (4.722) | 5.25 (3.202) | 6.25 (2.872)
  Eyes Closed: Maximum Change | 1.80 (2.588) | 2.00 (2.345) | -4.25 (2.630) | -6.25 (2.872)
  Eyes Opened: Baseline | 5.20 (5.404) | 4.60 (4.037) | 5.00 (3.830) | 6.25 (4.646)
  Eyes Opened: Maximum Change | 2.00 (3.240) | 1.80 (3.633) | -4.25 (3.304) | -6.25 (4.646)

5. Secondary Outcome: Duration of Mean Photosensitivity Response in Each of the 3 Eye Conditions (Eye Closure, Eyes Closed, and Eyes Open Condition) up to 8 Hours Postdose on Day 1 of Each Treatment Period
Description: Duration of mean photosensitivity response in each of the 3 eye conditions (eye closure, eyes closed, and eyes open condition) was determined from mean and mean change from baseline SPR data across participants. Duration of mean suppression was defined as the difference in hours between the onset of mean suppression and the end of mean suppression of photosensitivity across participants. The onset of mean suppression was defined as the first time point at which the mean SPR across participants was at least 3 units below the mean SPR at baseline. The end of mean suppression was defined as the last time (second time) with two successive reductions in mean SPR across participants of at least 3 units lower than the mean SPR at baseline. Photosensitivity response were essentially IPS assessments, is a form of visual stimulation, when the participants are flashed with light on their eyes intermittently at different hertz.
Time Frame: Baseline (30 minutes-2 hours) up to 8 hours postdose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Number; unit: hours
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
hours
  Eye Closure: Duration | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | 7 | 7
  Eyes Closed: Duration | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | 7 | 7
  Eyes Opened: Duration | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | NA — Duration of suppression cannot be determined because no suppression of photosensitivity by at least 3 units below the mean SPR at baseline was observed throughout the 8-hour assessment period on each day of treatment. | 7 | 7

6. Secondary Outcome: Number of Participants With Complete Suppression, Partial Response, and no Response of Standardized Photosensitivity Response (SPR) up to 8 Hours Postdose on Day 1 of Each Treatment Period
Description: Complete suppression, reduction (partial response), and no change (no response) of PPR will be measured. Complete suppression was defined as a SPR reduction to 0 over at least 1 time point for all three eye conditions. Partial response was defined as a reduction in SPR of at least 3 units from baseline for at least 3 time points, and no time points with at least 3 units of increase, in the most sensitive eye condition; without meeting the complete suppression definition. No response was defined as not meeting complete suppression or partial suppression definitions.
Time Frame: Baseline (30 minutes-2 hours) up to 8 hours postdose on Day 1 of each treatment period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
Participants
  Complete Suppression | 0 | 0 | 2 | 2
  Partial Response | 0 | 0 | 0 | 2
  No Response | 5 | 5 | 2 | 0

7. Secondary Outcome: Change From Baseline in Bond and Lader Visual Analogue Scales (BL-VAS) at 1, 2, 4, 6, and 8 Hours Post-dose in Each Treatment Period
Description: BL-VAS system was used to assess the extent of damage to the extrapyramidal system and the motor functions that it controls. The BL-VAS monitored the subjective mood of each participant on 16 mood scales. Participants were asked to indicate on the VAS scale ranging from 0 to 100 millimeter (mm) about how they felt at the moment the scale was administered (example, alert/drowsy; calm/excited; content/tensed). The individual responses from the 16 mood scales were then combined to make three subscales: a.) Anxiety, b.) Dysphoria, c.) sedation with each item ranges from 0 to 100 and higher scores indicated better condition.
Time Frame: Baseline (30 minutes-2 hours) and at 1,2,4,6 and 8 hours post-dose in each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
score on a scale
  Anxiety: Baseline | 29.42 (22.731) | 29.42 (22.731) | 24.33 (22.712) | 24.33 (22.712)
  Anxiety: Change at 1 hour post-dose | -7.36 (23.099) | -9.44 (19.550) | -0.37 (0.386) | -2.40 (3.382)
  Anxiety: Change at 2 hours post-dose | 2.84 (8.996) | -10.04 (20.028) | -1.05 (2.684) | 19.73 (42.748)
  Anxiety: Change at 4 hours post-dose | 2.82 (8.885) | -8.96 (18.512) | 0.10 (1.010) | -0.10 (4.017)
  Anxiety: Change at 6 hours post-dose | -0.72 (3.883) | -9.70 (21.895) | -0.87 (2.766) | -0.42 (4.452)
  Anxiety: Change at 8 hours post-dose | -0.72 (3.935) | 5.92 (43.792) | 18.78 (35.818) | -0.85 (3.171)
  Dysphoria: Baseline | 33.58 (23.032) | 33.58 (23.032) | 36.23 (25.703) | 36.23 (25.703)
  Dysphoria: Change at 1 hour post-dose | -4.44 (7.134) | -0.50 (6.536) | 0.50 (0.883) | 2.28 (4.110)
  Dysphoria: Change at 2 hours post-dose | 1.80 (3.616) | -1.62 (2.909) | 2.68 (3.886) | 3.30 (3.503)
  Dysphoria: Change at 4 hours post-dose | -0.26 (1.137) | -1.94 (3.889) | 2.47 (3.661) | 2.55 (3.486)
  Dysphoria: Change at 6 hours post-dose | -0.88 (3.397) | 1.56 (3.591) | 2.30 (3.866) | 0.02 (2.334)
  Dysphoria: Change at 8 hours post-dose | 0.30 (6.288) | -2.36 (3.965) | -0.30 (1.137) | -0.40 (1.337)
  Sedation: Baseline | 28.90 (18.748) | 28.90 (18.748) | 31.90 (20.215) | 31.90 (20.215)
  Sedation: Change at 1 hour post-dose | 4.36 (5.963) | 6.20 (4.933) | 6.45 (3.724) | 5.98 (4.131)
  Sedation: Change at 2 hours post-dose | 9.44 (9.060) | 7.23 (7.032) | 7.40 (4.291) | 8.18 (5.702)
  Sedation: Change at 4 hours post-dose | 5.50 (5.247) | 2.84 (6.993) | 11.55 (9.627) | 6.08 (4.219)
  Sedation: Change at 6 hours post-dose | 0.58 (2.567) | 2.70 (9.281) | 7.08 (4.424) | 10.30 (12.258)
  Sedation: Change at 8 hours post-dose | 1.08 (3.976) | 0.50 (6.615) | 2.38 (3.256) | 9.53 (9.466)

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Up to 28 days after the last dose of study treatment on Day 1 in Treatment Period 4 (approximately Day 71)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
Participants | 2 | 2 | 1 | 2

9. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: Up to 28 days after the last dose of study treatment on Day 1 in Treatment Period 4 (approximately Day 71)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Time Frame: Up to 28 days after the last dose of study treatment on Day 1 in Treatment Period 4 (approximately Day 71)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for E2082
Time Frame: Predose (within 2 hours prior to dosing) to 8 hours postdose on Day 1 of each treatment period
Population: The pharmacokinetic (PK) analysis set was the group of randomized participants who received at least 1 dose of study drug and have sufficient PK data to derive at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 4 | 4
nanogram per milliliter (ng/mL) | 100 (25.1) | 617 (30.3) | 851 (91.8)

12. Secondary Outcome: Tmax: Time to Reach Maximum Plasma Concentration (Cmax) for E2082
Time Frame: Predose (within 2 hours prior to dosing) to 8 hours postdose on Day 1 of each treatment period
Population: The PK analysis set was the group of randomized participants who received at least 1 dose of study drug and have sufficient PK data to derive at least 1 PK parameter.
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 4 | 4
hour | 3.93 [1.00 to 7.82] | 3.96 [3.90 to 4.00] | 3.99 [1.88 to 7.88]

13. Secondary Outcome: AUC (0-8h): Area Under the Plasma Concentration-time Curve From 0 to 8 Hours Post-dose for E2082
Time Frame: Predose (within 2 hours prior to dosing) to 8 hours postdose on Day 1 of each treatment period
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
Number analyzed (Participants) | 5 | 4 | 4
hour*nanogram per milliliter (h*ng/mL) | 633 (142) | 3990 (344) | 5750 (787)

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose of study treatment on Day 1 in Treatment Period 4 (approximately Day 71)
Arm/Group | Treatment A: Placebo | Treatment B: E2082 2.5 mg | Treatment C: E2082 25 mg | Open-label Treatment: E2082 40 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 2/5 | 1/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Placebo (N=5) | Treatment B: E2082 2.5 mg (N=5) | Treatment C: E2082 25 mg (N=4) | Open-label Treatment: E2082 40 mg (N=4)
Eye movement disorder (Eye disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Placebo (N=5) | Treatment B: E2082 2.5 mg (N=5) | Treatment C: E2082 25 mg (N=4) | Open-label Treatment: E2082 40 mg (N=4)
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 2
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Anger (Psychiatric disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to safety concerns from a phase 1 study (E2082-J081-001; NCT03402178) and preclinical animal toxicity testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT03686033/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03686033/SAP_001.pdf